CLINICAL TRIAL: NCT02359955
Title: Comparison of Masticatory Efficiency and EMG Activity Between Complete Denture With Zero-degree Teeth and Anatomic Teeth in Patients With Severely Resorbed Ridge
Brief Title: Comparison of Masticatory Efficiency Between Complete Denture With Zero-degree Teeth and Anatomic Teeth in Patients With Severely Resorbed Ridge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Haixin Qian (Other)
Responsible Party: Sponsor-Investigator, Haixin Qian, fellow, clinic research, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Organization: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 201395
Record Dates: First submitted 2015-01-23; First posted 2015-02-10 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Edentulous
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Zero-Degree Teeth, then Anatomic Teeth (Experimental): edentulous patients who were first treated with zero-degree teeth complete denture, then with anatomic teeth complete denture
  Interventions: Device: zero degree teeth; Device: anatomic teeth
- Anatomic Teeth, then Zero-Degree Teeth (Experimental): edentulous patients who were first treated with anatomic teeth complete denture, the with zero degree teeth complete denture
  Interventions: Device: zero degree teeth; Device: anatomic teeth

INTERVENTIONS:
Device: zero degree teeth — zero degree teeth complete denture was first prescribed to patients in group 1 while patients in group 2 were treated with anatomic teeth complete denture
Device: anatomic teeth — when anatomic teeth complete denture was prescribed to patients in group 1, patients in group 2 were treated with zero degree teeth complete denture

SUMMARY:
This study aims to evaluate masticatory efficiency of the zero-degree teeth complete denture in treatment of edentulous patients of severely resorbed ridge.Patients will be crossed over to be treated with zero-degree teeth complete denture and anatomic teeth complete denture. For each patient, the masticatory efficiency and electromyography with different denture will be recorded and analysis.

ELIGIBILITY:
Inclusion Criteria:

* complete edentulism for at least three months class Ⅳ ridge

Exclusion Criteria:

* neuromuscular dysfunction, psychiatric disorder,

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Estimated)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zero-degree Teeth, Then Anatomic Teeth | Anatomic Teeth, Then Zero-degree Teeth
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: edentulous patients who were first treated with zero-degree teeth complete denture, then with anatomic teeth complete denture
  zero degree teeth: zero degree teeth complete denture was first prescribed to patients in group 1 while patients in group 2 were treated with anatomic teeth complete denture
  anatomic teeth: when anatomic teeth complete denture was prescribed to patients in group 1, patients in group 2 were treated with zero degree teeth complete denture
- Group 2: edentulous patients who were first treated with anatomic teeth complete denture, the with zero degree teeth complete denture
  zero degree teeth: zero degree teeth complete denture was first prescribed to patients in group 1 while patients in group 2 were treated with anatomic teeth complete denture
  anatomic teeth: when anatomic teeth complete denture was prescribed to patients in group 1, patients in group 2 were treated with zero degree teeth complete denture
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (5.9) | 58.4 (5.29) | 58.65 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 5 | 9

OUTCOME MEASURES:

1. Secondary Outcome: Masticatory Efficiency Index
Description: the masticatory efficiency is tested after patient wears complete denture for three months,each patient was given 4 gram dry peanuts, chewed for 20 seconds, then spat in the receptacle and rinsed mouth residue. The peanut particles were diluted to 1000 ml with distilled water, stirred for 1 minutes and standing for 2 minutes to suspension. Absorbance values(av) were measured at the wavelength of 590nm in a spectrophotometer. The higher the masticatory efficiency, the smaller the peanut particles, then the higher the av value, vice versa. Value of av was used to represent masticatory efficiency. For each patient, the test was conducted three times, and the average value of av was taken as the final result. A lower masticatory efficiency index indicates larger peanut particle size observed.
Time Frame: three months
Measure: Mean (Standard Deviation); unit: index score
Groups:
- Group 1 Zero Degree Teeth: edentulous patients who were first treated with zero-degree teeth complete denture, then with anatomic teeth complete denture
- Group 2 Anatomic Teeth: edentulous patients who were first treated with anatomic teeth complete denture, the with zero degree teeth complete denture
Arm/Group | Group 1 Zero Degree Teeth | Group 2 Anatomic Teeth | Group 1 Anatomic Teeth | Group 2 Zero Degree Teeth
Number analyzed (Participants) | 10 | 10 | 10 | 10
index score | 0.327 (0.0714) | 0.334 (0.072) | 0.3364 (0.0996) | 0.329 (0.0862)

2. Primary Outcome: EMG (Masseters EMG Are Recorded After Patient Wears Complete Denture for Three Months)
Description: the masseters EMG are recorded after patient wears complete denture for three months,EMGs of masseters of 20 chewing strokes were recorded in term of value of amp and duration,amplitude is reported here as the average value from 20 chewing strokes in units of "microvolts".
Time Frame: three months
Measure: Mean (Standard Deviation); unit: microvolts
Groups:
- Amp Value of Right Masseter of Zero Degree Teeth: emg parameter of edentulous patients treated with zero-degree teeth complete denture
- Amp Value of Right Master of Anatomic Teeth: emg parameter of patients treated with anatomic teeth complete denture
Arm/Group | Amp Value of Right Masseter of Zero Degree Teeth | Amp Value of Left Masseter of Zero Degree Teeth | Amp Value of Right Master of Anatomic Teeth | Amp Value of Left Masseter of Anatomic Teeth
Number analyzed (Participants) | 20 | 20 | 20 | 20
microvolts | 0.72 (0.53) | 0.87 (0.49) | 1.07 (0.66) | 1.21 (1.00)

3. Primary Outcome: EMG (Masseters EMG Are Recorded After Patient Wears Complete Denture for Three Months)
Description: the masseters EMG are recorded after patient wears complete denture for three months,EMGs of masseters of 20 chewing strokes were recorded in term of value of amp and duration, duration here is reporteds the average value from 20 chewing strokes in units of "millisecond".
Time Frame: three month
Measure: Mean (Standard Deviation); unit: millisecond
Groups:
- Duration of Right Masseter of Zero Degree Teeth: emg parameter of patients treated with zero degree teeth
- Duration of Right Masster of Anatomic Teeth: emg parameter of patients treated with anatomic teeth complete denture
Arm/Group | Duration of Right Masseter of Zero Degree Teeth | Duration of Left Masseter of Zero Degree Teeth | Duration of Right Masster of Anatomic Teeth | Duration of Left Masseter of Anatomic Teeth
Number analyzed (Participants) | 20 | 20 | 20 | 20
millisecond | 247 (72) | 314 (82) | 306 (114) | 368 (102)

ADVERSE EVENTS:
Groups:
- Zero Degree Teeth,Then Anatomic Teeth: edentulous patients who were first treated with zero-degree teeth complete denture, then with anatomic teeth complete denture
Arm/Group | Zero Degree Teeth,Then Anatomic Teeth | Anatomic Teeth, Then Zero-degree Teeth
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes